CLINICAL TRIAL: NCT02691676
Title: Perioperative Fluid Therapy With Balanced Crystalloids: a Comparative Randomized Prospective Open Label Study
Brief Title: Perioperative Fluid Therapy With Balanced Crystalloids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Olomouc (Other)
Responsible Party: Principal Investigator, Radovan Uvizl, Radovan Uvizl, MD, Ph.D., University Hospital Olomouc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GV29125 16/14
Record Dates: First submitted 2016-02-10; First posted 2016-02-25 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Acid Base Imbalance
Keywords: crystalloids, fluid therapy, Plasmalyte, Ringerfundin
MeSH Terms: conditions — Acid-Base Imbalance | interventions — Plasmalyte A; Ringerfundin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plasmalyte (Experimental): Arm 1: Plasmalyte in 5% glucose infusion solution (PL), manufactured by Baxter Healthcare as slightly alkalizing (Na+ 140; K+ 5.0; Mg2+ 1.5; Cl- 98; acetate 27; gluconate 23)
  Interventions: Drug: Plasmalyte
- Ringerfundin (Active Comparator): Arm 2: Ringerfundin infusion solution (RF), manufactured by B. Braun as acid-base neutral (Na+ 145; K+ 4.0; Mg2+ 1.0; Ca2+ 2.5; Cl- 127; acetate 24; malate 5.0).
  Interventions: Drug: Ringerfundin

INTERVENTIONS:
Drug: Plasmalyte — Parenteral administration of Plasmalyte initiated immediately after collection of the first blood sample at 166 mL/hour. Thus, all patients received 1000 mL of infusion solution over 6 hours.
  Other Names: Plasmalyte (Baxter Healthcare)
  Arms: Plasmalyte
Drug: Ringerfundin — Parenteral administration of Ringerfundin initiated immediately after collection of the first blood sample at 166 mL/hour. Thus, all patients received 1000 mL of infusion solution over 6 hours.
  Other Names: Ringerfundin (B. Braun)
  Arms: Ringerfundin

SUMMARY:
Introduction: The strategy of perioperative fluid therapy has an important impact not only on the circulating volume and perfusion of organs and tissues but also on the patient's internal environment. The study aimed at comparing the effects of perioperatively administered balanced crystalloid infusion solutions containing different amounts of metabolizable anions on homeostasis.

Methods: In the prospective randomized study, patients were assigned to Plasmalyte (PL) and Ringerfundin (RF) Groups after their postoperative transfer to an intensive care unit (ICU). The infusion solutions were parenterally administered at 1000 mL/6 hours. Arterialized capillary blood was sampled at the time of transfer to the ICU (Time 0), and again at 2 hours and 6 hours from Time 0. The collected blood was tested for blood gas parameters using the Astrup method.

DETAILED DESCRIPTION:
Study design

The study was designed as a single-center, randomized, prospective study and approved by the University Hospital Olomouc and Faculty of Medicine and Dentistry, Palacky University Olomouc ethics committee. It comprised patients over 18 years of age undergoing surgery at the hospital's Department of Surgery I and subsequently placed in an ICU bed. As there were no limitations concerning the type of procedures, these involved a wide range of abdominal and thoracic surgeries; however, all of them were elective procedures. No patients were critically ill, being classified as ASA III or less.

Sample collection and processing To determine the present status of the internal environment, arterialized capillary blood was drawn from the fingertip at the time of patients' transfer from the operating room to the ICU (Time 0), and again at 2 hours and 6 hours from Time 0. The collected blood was tested in the laboratory using the Astrup method to measure the following parameters: pH, BE, actual bicarbonate (aBi), standard bicarbonate (sBi), partial pressure of oxygen (pO2) and carbon dioxide (pCO2). The obtained values were entered into a table and statistically analyzed. Both patients groups were adjusted for age and length of surgery to allow their comparison.

Infusion solutions

The following infusion solutions were parenterally administered using a central or, more frequently, peripheral venous catheter:

1. Plasmalyte in 5% glucose infusion solution (PL), manufactured by Baxter Healthcare as slightly alkalizing (Na+ 140; K+ 5.0; Mg2+ 1.5; Cl- 98; acetate 27; gluconate 23) and
2. Ringerfundin infusion solution (RF), manufactured by B. Braun as acid-base neutral (Na+ 145; K+ 4.0; Mg2+ 1.0; Ca2+ 2.5; Cl- 127; acetate 24; malate 5.0).

At the time of their transfer to the ICU, patients were randomized into PL and RF Groups. Parenteral administration of the two solutions was initiated immediately after collection of the first blood sample at 166 mL/hour. Thus, all patients received 1000 mL of infusion solution over 6 hours. Patients requiring more rapid fluid replacement due to postoperative hypovolemia were excluded from the study. Patients were routinely rewarmed with a warm air blanket and received humidified oxygen via a face mask or, in case of good oxygenation, via a nasal cannula.

ELIGIBILITY:
Inclusion Criteria:

* age 18+
* elective surgery procedures

Exclusion Criteria:

* critically ill, being classified as ASA III or less
* surgery longer than 6 hrs
* hypersensitivity to PL or RF
* requiring more rapid fluid replacement (than 1000 ml/6 hrs) due to postoperative hypovolemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with significant acid basic disturbances related to balanced alkalizing as compared with a balanced pH-neutral crystalloids. | 6 hours
  The internal environment status is assessed at the time of patients' transfer from the operating room to the ICU (Time 0), and again at 6 hours from Time 0. Outcome over a longer period of time is not rated.

CONTACTS AND LOCATIONS:
Overall Officials: Radovan Uvizl, Principal Investigator — University Hospital Olomouc

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zadak Z, Hyspler R, Hronek M, Ticha A. The energetic and metabolic effect of Ringerfundin (B. Braun) infusion and comparison with Plasma-Lyte (Baxter) in healthy volunteers. Acta Medica (Hradec Kralove). 2010;53(3):131-7. doi: 10.14712/18059694.2016.72. PMID 21171525
- [Background] Kirkendol PL, Starrs J, Gonzalez FM. The effects of acetate, lactate, succinate and gluconate on plasma pH and electrolytes in dogs. Trans Am Soc Artif Intern Organs. 1980;26:323-7. No abstract available. PMID 7245507
- [Background] Zavorsky GS, Cao J, Mayo NE, Gabbay R, Murias JM. Arterial versus capillary blood gases: a meta-analysis. Respir Physiol Neurobiol. 2007 Mar 15;155(3):268-79. doi: 10.1016/j.resp.2006.07.002. Epub 2006 Aug 17. PMID 16919507
- [Background] Lowell JA, Schifferdecker C, Driscoll DF, Benotti PN, Bistrian BR. Postoperative fluid overload: not a benign problem. Crit Care Med. 1990 Jul;18(7):728-33. doi: 10.1097/00003246-199007000-00010. PMID 2364713
- [Background] Holte K, Jensen P, Kehlet H. Physiologic effects of intravenous fluid administration in healthy volunteers. Anesth Analg. 2003 May;96(5):1504-1509. doi: 10.1213/01.ANE.0000055820.56129.EE. PMID 12707158
- [Background] Bouchard JE, Mehta RL. Fluid balance issues in the critically ill patient. Contrib Nephrol. 2010;164:69-78. doi: 10.1159/000313722. Epub 2010 Apr 20. PMID 20427995
- [Background] Simmons RS, Berdine GG, Seidenfeld JJ, Prihoda TJ, Harris GD, Smith JD, Gilbert TJ, Mota E, Johanson WG Jr. Fluid balance and the adult respiratory distress syndrome. Am Rev Respir Dis. 1987 Apr;135(4):924-9. doi: 10.1164/arrd.1987.135.4.924. PMID 3565940
- [Background] Rahbari NN, Zimmermann JB, Schmidt T, Koch M, Weigand MA, Weitz J. Meta-analysis of standard, restrictive and supplemental fluid administration in colorectal surgery. Br J Surg. 2009 Apr;96(4):331-41. doi: 10.1002/bjs.6552. PMID 19283742
- [Background] Kocian P, Neumann J, Majtan P, Hoch J. [Fluid therapy and surgical outcomes after low anterior resection]. Rozhl Chir. 2014 Sep;93(9):463-7. Czech. PMID 25301345
- [Background] Brandstrup B. Fluid therapy for the surgical patient. Best Pract Res Clin Anaesthesiol. 2006 Jun;20(2):265-83. doi: 10.1016/j.bpa.2005.10.007. PMID 16850777
- [Background] Nisanevich V, Felsenstein I, Almogy G, Weissman C, Einav S, Matot I. Effect of intraoperative fluid management on outcome after intraabdominal surgery. Anesthesiology. 2005 Jul;103(1):25-32. doi: 10.1097/00000542-200507000-00008. PMID 15983453
- [Background] Holte K, Klarskov B, Christensen DS, Lund C, Nielsen KG, Bie P, Kehlet H. Liberal versus restrictive fluid administration to improve recovery after laparoscopic cholecystectomy: a randomized, double-blind study. Ann Surg. 2004 Nov;240(5):892-9. doi: 10.1097/01.sla.0000143269.96649.3b. PMID 15492573
- [Result] Chowdhury AH, Cox EF, Francis ST, Lobo DN. A randomized, controlled, double-blind crossover study on the effects of 1-L infusions of 6% hydroxyethyl starch suspended in 0.9% saline (voluven) and a balanced solution (Plasma Volume Redibag) on blood volume, renal blood flow velocity, and renal cortical tissue perfusion in healthy volunteers. Ann Surg. 2014 May;259(5):881-7. doi: 10.1097/SLA.0000000000000324. PMID 24253140